CLINICAL TRIAL: NCT00024401
Title: Phase II Open-Label Study of Taxoperxin (DHA-Paclitacel) Injection by 2-Hour Intravenous Infusion in Patients With Metastatic Cancer of the Colon/Rectum
Brief Title: DHA-Paclitaxel in Treating Patients With Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Theradex (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068929; THERADEX-P01-00-01; ABCCC-010505; PROTARGA-P01-00-01
Record Dates: First submitted 2001-09-13; First posted 2004-01-15 (Estimated); Last update posted 2008-07-24 (Estimated); Status verified 2002-06

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — docosahexaenoyl-paclitaxel

INTERVENTIONS:
Drug: DHA-paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of DHA-paclitaxel in treating patients who have metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the objective tumor response rate, duration of response, and time to disease progression in patients with metastatic colorectal cancer treated with DHA-paclitaxel. II. Determine the overall survival of patients treated with this drug. III. Determine the toxicity profile of this drug in these patients. IV. Assess the quality of life of patients treated with this drug.

OUTLINE: This is a multicenter study. Patients receive DHA-paclitaxel IV over 2 hours on day 1. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity. Quality of life is assessed at baseline, every 2 courses, and at end of study treatment. Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 18-50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed cancer of the colon or rectum Clinical evidence of metastatic disease Failed 1 prior chemotherapy regimen for metastatic disease Measurable disease No known or clinical evidence of CNS metastasis

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-1 Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 times upper limit of normal (ULN) SGOT or SGPT no greater than 2.5 times ULN Renal: Creatinine no greater than 1.5 times ULN Cardiovascular: No uncontrolled ventricular arrhythmia No myocardial infarction within the past 3 months No superior vena cava syndrome Neurologic: No peripheral neuropathy greater than grade 1 No uncontrolled major seizure disorder No spinal cord compression Other: No unstable or serious concurrent medical condition No concurrent serious infection requiring parenteral therapy No other prior malignancy except: Curatively treated nonmelanoma skin cancer or carcinoma in situ of the cervix OR Other cancer curatively treated with surgery alone that has not recurred for more than 5 years No psychiatric disorder that would preclude study Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception during and for 6 months after study

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent immunotherapy Chemotherapy: See Disease Characteristics No more than 1 prior chemotherapy regimen for metastatic disease No prior taxanes At least 28 days since prior chemotherapy and recovered No other concurrent chemotherapy Endocrine therapy: No concurrent hormonal therapy Radiotherapy: At least 28 days since prior large-field radiotherapy and recovered No concurrent radiotherapy Surgery: At least 14 days since prior major surgery and recovered

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-05

CONTACTS AND LOCATIONS:
Overall Officials: Ross C. Donehower, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (6):
- United States (6):
  - Arizona Oncology Associates, Tucson, Arizona
  - Veterans Affairs Medical Center - Washington, DC, Washington D.C., District of Columbia
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey